CLINICAL TRIAL: NCT02004132
Title: A Phase 1, Single-Dose Study to Evaluate Testosterone on Clothing After Axiron® Use in Healthy Male Subjects
Brief Title: A Study of Axiron® in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15281; I5E-EW-TSBE (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-12-03; First posted 2013-12-06 (Estimated); Results first posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Testosterone Propionate; Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Axiron (Experimental): Axiron administered topically via metered dose pump to each underarm on Day 1
  Interventions: Drug: Axiron

INTERVENTIONS:
Drug: Axiron — Solution administered topically using pump and applicator
  Other Names: LY900011; Testosterone

SUMMARY:
The study involves application of Axiron to each underarm. The study will evaluate the transfer of testosterone from underarms to the clothing items that the participant is wearing and other fabric items washed with participant's' clothes. The study is approximately 6 days, not including screening. Screening is required within 28 days prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males, as determined by medical history and physical examination, or males who have been on stable medication for at least 1 month and have no significant clinical conditions.
* Agree to use a reliable method of birth control (for example: condom or vasectomy) during the study and for 3 months following the Axiron dose
* Have clinical laboratory test results within the normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures
* Have given written informed consent approved by Lilly and the ethical review board (ERB) governing the site

Exclusion Criteria:

* Are currently enrolled in a clinical trial involving an investigational product or off-label use of a drug or device, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Are participants who have previously completed or withdrawn from this study or any other study investigating Axiron in the past 3 months
* Have known allergies to testosterone solution, related compounds, or any components of the formulation, or history of significant atopy
* Have an abnormality in the 12-lead electrocardiogram (ECG) that, in the opinion of the investigator, increases the risks associated with participating in the study
* Have an abnormal blood pressure as determined by the investigator
* Have a history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders constituting a risk when taking the study medication or that could interfere with the interpretation of the data
* Have had lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen
* Use of any topical testosterone replacement therapy within the 3 months prior to study entry through study discharge, except for use of Axiron as directed by study procedures
* Use of parenteral testosterone replacement (testosterone enthanate, testosterone cypionate) within the 30 days prior to screening. Use of long acting intramuscular testosterone undecanoate 6 months prior to screening, or use of testosterone pellets 12 months prior to screening
* Have a dermatologic condition in the underarm area that might be exacerbated by topical testosterone replacement therapy, in the opinion of the investigator
* In the opinion of the investigator or sponsor, are unsuitable for inclusion in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daytona Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Axiron 120 mg: Single 120 milligrams (mg) total dose given to participants as two 1.5 milliliters (mL) topical applications to each underarm (60 mg per underarm) in the morning on Day 1 using a pump.
Period: Overall Study
Arm/Group | Axiron 120 mg
Started | 12
Received Study Drug | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received a dose of study drug.
Arm/Group | Axiron 120 mg
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Amount of Testosterone on T-shirts
Description: This is a summary of the amounts of testosterone measured on a 10 centimeters (cm) × 10 cm of material excised from the underarm area of participant's unwashed t-shirt halves.
Time Frame: 12 hours after application of study drug
Population: Full analysis set (FAS). Data from all enrolled participants completing the study.
Measure: Mean (Standard Deviation); unit: micrograms (µg)
Arm/Group | Axiron 120 mg
Number analyzed (Participants) | 12
micrograms (µg) | 7603 (2790)

2. Secondary Outcome: Amount of Testosterone Following Laundering
Description: This is a summary of the amounts of testosterone measured on a 10 cm × 10 cm of material excised from the underarm area of washed t-shirt halves following laundering in a standard washing machine.
Time Frame: 12 hours after application of study drug
Population: FAS. Data from all enrolled participants completing the study.
Measure: Mean (Standard Deviation); unit: µg
Arm/Group | Axiron 120 mg
Number analyzed (Participants) | 12
µg | 260 (407)

3. Secondary Outcome: Amount of Testosterone on Unworn Textiles Laundered With the Testosterone Exposed T-shirts
Description: This is a summary of the amounts of testosterone measured on unworn textile items washed with t-shirt halves exposed to testosterone in a standard washing machine. Total amounts of testosterone on each laundered item other than the t-shirt halves was calculated based on the weight of the fabric sample analyzed and the total weight of the item, assuming a uniform distribution of testosterone across each item as:
  (weight of laundered item / weight of laundered sample) x amount of testosterone on laundered sample.
Time Frame: 12 hours after application of study drug
Population: FAS. Data from all enrolled participants completing the study.
Measure: Mean (Standard Deviation); unit: µg
Arm/Group | Axiron 120 mg
Number analyzed (Participants) | 12
µg
  Bleached Cotton Terry Cloth | 308 (71.9)
  Wool Jersey Knit Fabric | 122 (23.8)
  56/44 Cotton/Linen | 441 (70.8)
  Texturized Dacron 56T Double | 68.7 (21.0)
  87/13 Nylon/Lycra Knit | 10402 (1408)

ADVERSE EVENTS:
Time Frame: Randomization up to 9 days follow-up
Description: Events deemed to be serious adverse events (SAEs) by the Investigator as related to study drug administration were collected during the study and up to 9 days following study drug administration.
Arm/Group | Axiron 120 mg
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Axiron 120 mg (N=12)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days